CLINICAL TRIAL: NCT05989659
Title: Transitioning Patients with Advanced Chronic Kidney Disease to Home or In-center Dialysis: Understanding the Experience and Quality of Life for Patients and Their Caregivers
Brief Title: Transitioning to Home or In-center Dialysis
Acronym: TRANSIT-CARE
Status: Recruiting | Type: Observational
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The Kidney Foundation of Canada (Other)
Responsible Party: Sponsor
Other Study IDs: 2022_2973
Record Dates: First submitted 2023-07-28; First posted 2023-08-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Chronic Kidney Diseases
Keywords: Chronic Kidney Disease; Quality of Life; Frailty; Home Dialysis; Peritoneal Dialysis; Home Hemodialysis; Hemodialysis; Mixed Methods
MeSH Terms: conditions — Renal Insufficiency, Chronic; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Patient - Home Dialysis: Patients transitioning to home dialysis
  Interventions: Other: Exposure: Home dialysis or facility-hemodialysis
- Patient - Facility Hemodialysis: Patients transitioning to facility hemodialysis
  Interventions: Other: Exposure: Home dialysis or facility-hemodialysis
- Caregivers - Home dialysis: Caregivers of patients transitioning to home dialysis
  Interventions: Other: Exposure: Home dialysis or facility-hemodialysis
- Caregivers - Facility Hemodialysis: Caregivers of patients transitioning to facility hemodialysis
  Interventions: Other: Exposure: Home dialysis or facility-hemodialysis

INTERVENTIONS:
Other: Exposure: Home dialysis or facility-hemodialysis — Initiation of dialysis with home dialysis (peritoneal dialysis or home hemodialysis) or facility-hemodialysis

SUMMARY:
For people with advanced kidney disease, deciding which type of dialysis is best can be challenging. Studies have shown that quality of life is very important to patients. It is thought that the quality of life of people receiving their dialysis at home may be better than the one of people receiving dialysis in a hospital. However, how the start of dialysis changes the quality of life of people who choose home dialysis in comparison to people choosing dialysis in a hospital is still unknown.

TRANSIT-CARE is a prospective mixed methods study following adult with advanced kidney disease who progress to dialysis and receive home or hospital-based dialysis. This study aims to examine the trajectory and change in patients' quality of life and their frailty status (health, mobility and function) before start of dialysis and up to 12-month after start. Differences between people doing home dialysis and hospital-based dialysis will be assesses taking into account people's characteristics including their gender and socio-demographics characteristics. The study will include questionnaires to measure quality of life and tools to evaluate frailty. Additionally, semi-structured interviews will be done with a diverse group of patients and caregivers before and after the initiation of dialysis to better understand their experience of transitioning to dialysis.

DETAILED DESCRIPTION:
Home dialysis has been encouraged due to its clinical benefits and lower costs, leading to increased use in recent years, even among patients with a high comorbidity burden and frailty severity. Health-related quality of life (HRQoL) is reduced in patients receiving dialysis, although patients treated with home dialysis may have relatively better patient-reported outcome measures (PROMs), than those on in-center dialysis. As the home dialysis population expands to include patients with a high frailty severity, it is unknown if these benefits are preserved. More importantly, data lacks on how the transition to home or in-center dialysis is experienced by patients and caregivers and whether changes in HRQoL and frailty impact this experience.

Objectives

1. Determine and compare the trajectory of HRQoL, frailty and caregiver burden during the chronic kidney disease (CKD)-to-dialysis transition. (QUANTI)
2. Examine the experience of participants during their progression from CKD to dialysis. (QUALI)
3. Understand how HRQoL, frailty, and dialysis modality influence patients' and caregivers' experience of transition. (QUANTI+QUALI)

Design and Research Plan TRANSIT-CARE is a 5-year multicenter mixed-methods study of patients with advanced CKD and their caregivers across 12 Canadian centers, with active patient-partner engagement.

QUANTITATIVE Participant will be followed every 3-months (from estimated glomerular filtration rate [eGFR] <12 mL/min/1.73m2) and up to 12-month after dialysis start (4-week, 3-, 6-,12-month).

Target recruitment: 420 patients / 165 caregivers. Dialysis modality will be defined as the chosen modality at baseline visit, and dichotomized as home dialysis (peritoneal or home hemodialysis) and in-center dialysis.

Changes in PROMs and frailty will be assessed using multivariable mixed linear spline regression analysis with each measure used as a continuous variable adjusted for baseline scores, chosen dialysis modality (exposure), dialysis start (time-dependent variable) and prespecified potential confounders.

QUALITATIVE Semi-structured interviews will be conducted with 30 patients and 30 caregivers (from three centers) before and after dialysis initiation.

Thematic analysis will be used to identify patient and caregiver perceptions of home and in-center dialysis, their reactions to dialysis initiation (e.g., feelings of empowerment or loss, life disruption) and perceived burden for caregivers.

Data integration Data from the qualitative and quantitative components will be integrated at time of analysis using tables and joint displays.

ELIGIBILITY:
Inclusion Criteria:

1. Adults followed in advanced CKD clinic,
2. estimated glomerular filtration rate (eGFR) <12 mL/min/1.73m2 103,
3. Have chosen their dialysis modality,
4. Understand English or French.

Exclusion Criteria:

1. Orientation toward conservative treatment,
2. Planned kidney transplantation < 6 months,
3. Unable to provide consent due to severe cognitive or psychiatric disease,
4. Previous treatment with dialysis > 3 months,
5. Life expectancy < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults followed in advanced chronic kidney disease clinics and their caregivers will be recruited from 12 academic centers across Canada
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Kidney Disease Quality of Life - 36 (KDQOL-36) - Patients | From study inclusion until 12-months after dialysis start.
  Scale from 0-100 (0=poor , 100 = excellent )
Change in 'ZARIT' burden Interview (ZBI) - Caregivers | From study inclusion until 12-months after dialysis start.
  Scale 0-88 (0=no/little burden, 88 = severe burden)

SECONDARY OUTCOMES:
Change in Fried Frailty phenotype | From study inclusion until 12-months after dialysis start.
  5 components (slowness, weakness, weight loss, low physical activity, exhaustion) with classification as no-frail, pre-frail or frail
Change in Clinical Frailty Scale | From study inclusion until 12-months after dialysis start.
  Scale 1 (very fit) to 9 (terminally ill)
Change in Hospital Anxiety and Depression - Patients | From study inclusion until 12-months after dialysis start.
  14-item scale (7 anxiety, 7 depression) with score ≥8 used as cut-off for increased risk of depression and anxiety
Change in Short-form (SF)-36 - Caregivers | From study inclusion until 12-months after dialysis start.
  Scale from 0-100 (0=poor , 100 = excellent )

OTHER OUTCOMES:
Semi-structured interviews with patients and caregivers | First interview between study start and dialysis initiation / Second interview between dialysis start and up to 12-month after dialysis start.
  2 interviews with patients and caregivers

CONTACTS AND LOCATIONS:
Overall Officials: Annie-Claire Nadeau-Fredette, MD, Principal Investigator — CIUSSS de l'Est-de-l'Ile-de-Montréal
Locations (1):
- Hôpital Maisonneuve-Rosemont, Montreal, Quebec, Canada